CLINICAL TRIAL: NCT07256106
Title: Evaluation of The Occlusion and Dis-Occlusion Time in Mandibular Single Overdentures Supported by Conventional Versus Mini- Dental Implants; A Parallel Blinded Randomized Clinical Trial
Brief Title: Occlusion and Dis-Occlusion Time in Mandibular Overdentures Supported by Conventional Versus Mini- Dental Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Abdelfatah, Associate professor , faculty of dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECIR072505
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Dental Implant; Edentulous Mouth
Keywords: occlusion time; disocclusion time
MeSH Terms: conditions — Mouth, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT) with parallel assignment of the participants in two groups in ratio 1:1. Randomization will be guided by a computer-generated list. Both groups will be placed in twenty eight numbered closed opaque sealed envelopes according to the computer generated list of random numbers and an envelope will be allocated to each patient. For allocation concealment, one of the postgraduate students who will be the only one to know the key so that the authors and the patients won't know in which group the patient will be. Afterwards, the authors will be informed by the randomization to be tabulated.
Who Masked: Outcomes Assessor
Masking Description: Masking of the outcome assessor the one responsible for measuring the occlusion/dis occlusion time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional implant supported mandibular overdenture (Active Comparator): Group CI patients will be rehabilitated with mandibular overdentures retained by two immediately loaded conventional implants inserted in the inter-foraminal region.
  Interventions: Procedure: conventional dental implant
- mini-implant supported mandibular overdenture (Experimental): Group MI patients will be rehabilitated with single mandibular overdentures retained by four immediately loaded mini implants inserted in the inter-foraminal region.
  Interventions: Procedure: mini dental implant

INTERVENTIONS:
Procedure: mini dental implant — For group MI patient, four screw type one piece mini dental implants will be inserted in the predetermined implant sites in the symphesial region. The position of the two distal implants will be marked 6 mm mesial to each mental foramen. The position of the other two implants will be marked equidistant from the distal implants with and at least 5 mm apart
  Arms: mini-implant supported mandibular overdenture
Procedure: conventional dental implant — For group CI patient, two screw type conventional implants will be inserted in the symphesial region.
  Arms: conventional implant supported mandibular overdenture

SUMMARY:
The aim of the study will be comparing between the occlusion and disocclusion time in mandibular single overdenture supported with immediately loaded two conventional implants versus immediately loaded four mini-implants.

Research question Is there a difference in occlusion and disocclusion time between two mandibular single dentures, one supported by immediately loaded two conventional implants and the second one supported by immediately loaded four mini-implants? Primary outcome: occlusion and disocclusion time Secondary outcome: Kapur index The null hypothesis is that there is no difference between both treatment modalities on occlusion and disocclusion time.

DETAILED DESCRIPTION:
Twenty eight patients will be selected to share in this study from the outpatient clinic of Prosthodontics Department, Faculty of Dentistry, Ain-Shams University.

Sample size was calculated according to these values producing a minimal sample size of Twenty eight patients being enough to find such a difference. The size was determined in the light of the study " Computerized occlusal analysis of mini-dental implant-retained mandibular overdentures: A 1-year prospective clinical study " 34 with alpha error probability of 0.05, 1-beta error probability , power of 0.8 and drop out ratio 5%.

The inclusion criteria will be patients with completely edentulous lower ridges and fully dentate or partially dentate maxillary arch restored with fixed restoration, exhibiting enough inter-arch space to allow for prosthetic rehabilitation with lower implant-retained overdentures and have good oral hygiene and motivation. The excluded patients will be patients with major systemic diseases that may affect osseointegration as uncontrolled diabetes mellitus, pregnancy, patients under bisphosphonate treatment.

The patients will make a complete oral and radiographic examination before inclusion in this study.

For allocation concealment, one of the postgraduate students who will be the only one to know the key so that the authors and the patients won't know in which group the patient will be. Afterwards, the authors will be informed by the randomization to be tabulated.

Ethical approval will be granted by the research ethics committee in the Faculty of Dentistry Ain Shams University (FDASUREC). All patients will be informed in details about the nature of the investigation and the aim of the study. Patients' data will be kept safe and confidential to protect the security and privacy of the patient information. All participants will be given notice about their privacy and their rights.

The patients will be divided into two equal groups; group (CI) and group (MI). Group CI patients will be rehabilitated with mandibular overdentures retained by two immediately loaded conventional implants inserted in the inter-foraminal region.

Group MI patients will be rehabilitated with single mandibular overdentures retained by four immediately loaded mini implants inserted in the inter-foraminal region.

During the first appointment, medical history, clinical and radiological evaluation will be recorded to verify the eligibility of each subject. To assess the residual bone anatomy, a CBCT scan will be performed according to the manufacturer's instructions with a proper field-of-view size to include both the upper and lower jaw. All patients were rehabilitated with complete single mandibular dentures prior to implant insertion. A radiopaque markers will be added to the patient's mandibular denture to make a radiographic stent. For each patient in both groups a CBCT will be made while wearing the radiographic stent.

Surgical procedures:

All surgical procedures will be performed under local anesthesia on an outpatient basis by the same surgical team.

For group CI patient, two screw type conventional implants will be inserted in the symphesial region. Crestal incision extending about 5 mm distal to each proposed implant sites will be made. A full thickness mucoperiosteal flap will be reflected exposing the bone in the proposed area.

A round bur will be used to mark the implant sites guided by the surgical stent. Preparation of implant site will start with the pilot drill placed parallel to the midline in both implant sites. Two paralleling tools will be used to check parallelism. The osteotomy preparation will be continued until the final drill. Implants will be threaded in place and the mucoperiosteal flap will be repositioned and sutured.

For group MI patient, four screw type one piece mini dental implants will be inserted in the predetermined implant sites in the symphesial region. The position of the two distal implants will be marked 6 mm mesial to each mental foramen. The position of the other two implants will be marked equidistant from the distal implants with and at least 5 mm apart.

At the marked implant site, Cortical drill will be used to penetrate cortical bone. A pilot drill will be used to drill bone up and down in a vertical direction until the desired length reached. The implant will be picked up from the sterile vial and directly inserted into the prepared site.

Post-surgical procedures:

After the surgery, areas opposing to the inserted implants will be marked on the fitting surfaces of the mandibular single denture. Abrasive stone will be used to relieve the marked areas and create enough space for the metal housing, The metal housings will be seated on the implant heads. The denture will be placed in the patient's mouth to check and ensure complete seating and proper inter-cuspal relation. Auto-polymerized dough acrylic resin will be mixed and added to the relieved areas and the denture will be reseated inside the patient's mouth. Patients will be instructed to close in centric until complete polymerization take place. The lower single denture will be removed from the patient's mouth with the metal housings in the fitting surface. The excess acrylic resin will be removed.

Method of evaluation:

Occlusal parameters: occlusion time (OT) and disocclusion time (DT) will be recorded for each patient. The patient will be asked to close on sensor in centric occlusion holding their teeth together for 1 to 3 seconds then start right eccentric movement until disoccluding their teeth. The patient will then be asked to close on sensor in centric occlusion holding their teeth together for 1 to 3 seconds then start left eccentric movement until disoccluding their teeth. This will be repeated 4 times for the right excursion (DT-right) and 4 times for the left excursion (DT-left). OT, DT-right, and DT-left were then calculated by taking the averages of the recordings.

The retention and stability of the conventional dentures will be assessed intra-orally by a single experienced examiner using the modified Kapur criteria (Olshan modification).

ELIGIBILITY:
Inclusion Criteria:

* patients with completely edentulous mandibular ridges and fully dentate or partially dentate maxillary arch restored with fixed restoration,

  * enough inter-arch space to allow for prosthetic rehabilitation with lower implant-retained overdentures
  * good oral hygiene and motivation.

Exclusion Criteria:

* The excluded patients will be patients with major systemic diseases that may affect osseointegration as uncontrolled diabetes mellitus, pregnancy, patients under bisphosphonate treatment.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
occlusion/dis occlusion time | 1 year
  Occlusal parameters: occlusion time (OT) and disocclusion time (DT) will be recorded for each patient. The patient will be asked to close on sensor in centric occlusion holding their teeth together for 1 to 3 seconds then start right eccentric movement until disoccluding their teeth. This will be repeated 4 times for the right excursion (DT-right) and 4 times for the left excursion (DT-left). OT, DT-right, and DT-left were then calculated by taking the averages of the recordings.

SECONDARY OUTCOMES:
denture stability | 1 year
  stability of the over dentures will be assessed intra-orally by a single experienced examiner using the modified Kapur criteria (Olshan modification).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed, MD, Principal Investigator — Faculty of dentistry, ain shams university
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt